CLINICAL TRIAL: NCT02779686
Title: PIIR Study: Comparison of Genetic Tests for Age-Related Macular Degeneration
Acronym: PIIR
Status: Terminated | Type: Observational
Why Stopped: Investigator left institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 1200081
Record Dates: First submitted 2016-05-13; First posted 2016-05-20 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Age-Related Macular Degeneration (ARMD)
Keywords: Macular Degeneration; Genetic testing; Age-Related Macular degeneration; Age-Related Maculopathies
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ARMD Free: Patient free of ARMD on clinical examination
- ARMD Positive: Patients with evidence of ARMD on clinical examination

SUMMARY:
This study is being conducted to compare two different genetic tests developed to determine an individuals risk of developing serious vision threatening complications from age-related macular degeneration (ARMD).

DETAILED DESCRIPTION:
There are currently two different genetic tests that have been developed for this purpose. They both look at specific DNA components to determine the risk. Participants in the study will be over the age of 60 years and caucasian as this is the population of people in which these tests have been validated. Each participant will have the study explained to them and then will be asked to sign the informed consent document if they agree to participate. They will have a dilated exam of their eyes along with photographs taken of the retina. If their doctor sees that it is necessary they will also have a special scan or a special angiogram of their eyes to look at their retina in more detail. For the genetic testing a member of the research team will use two swabs from each of the genetic companies to gently scrap some cells from the inside of the cheek. These cells will be sent to each respective lab for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian race
* Age >/= 60 years
* Patient's written informed consent
* Ability to comply with the protocol procedures

Exclusion Criteria:

* Race other than Caucasian
* Age < 60 years
* Macular or retinal pathology other than ARMD
* Known hypersensitivity to any drug included in the treatment protocol
* Any other severe clinical condition that in the judgment of the local investigator would place the patient at undue risk or interfere with the study completion
* Prisoners

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caucasian patients over the age of 60
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Risk score from RetnaGene | Day 1
  Risk score assigned after genetic analysis of a buccal swab by the RetnaGene (Sequenom) genetic test.
Risk score from Macula Risk | Day 1
  Risk score assigned after genetic analysis of a buccal swab by the Macula Risk genetic test.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Holekamp, MD, Principal Investigator — Pepose Vision Institute; Mathew MacCumber, MD, PhD, Principal Investigator — Rush University Medical Center; Arghavan Almony, MD, Principal Investigator — University of Missouri-Columbia
Locations (3):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - Pepose Vision Institute, Chesterfield, Missouri
  - University of Missouri-Columbia, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seddon JM, Reynolds R, Maller J, Fagerness JA, Daly MJ, Rosner B. Prediction model for prevalence and incidence of advanced age-related macular degeneration based on genetic, demographic, and environmental variables. Invest Ophthalmol Vis Sci. 2009 May;50(5):2044-53. doi: 10.1167/iovs.08-3064. Epub 2008 Dec 30. PMID 19117936
- [Background] Hageman GS, Gehrs K, Lejnine S, Bansal AT, Deangelis MM, Guymer RH, Baird PN, Allikmets R, Deciu C, Oeth P, Perlee LT. Clinical validation of a genetic model to estimate the risk of developing choroidal neovascular age-related macular degeneration. Hum Genomics. 2011 Jul;5(5):420-40. doi: 10.1186/1479-7364-5-5-420. PMID 21807600
- [Background] Zanke B, Hawken S, Carter R, Chow D. A genetic approach to stratification of risk for age-related macular degeneration. Can J Ophthalmol. 2010 Feb;45(1):22-7. doi: 10.3129/i09-209. PMID 20130705
- See also: RetnaGene product/test information — http://www.sequenom.com
- See also: Macula Risk product/test information — http://www.macularisk.com